CLINICAL TRIAL: NCT01441869
Title: Bioequivalence Study of the Fixed-dose Combination of Saxagliptin/Metformin XR Tablets Relative to Saxagliptin (Onglyza� ) Tablets and Australia-sourced Diabex XR Tablets Coadministered to Healthy Subjects in the Fed State During Steady-state Administration
Brief Title: Study in Healthy Subjects to Measure Amount of Drug in Blood After Dosing With Different Saxagliptin / Metformin Produc
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D1681C00004
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Bioequivalence, Log-transformed AUCss and Cmax,ss Values for Saxagliptin and Metformin
Keywords: Phase 1, Healthy male volunteers, pharmacokinetics, saxagliptin/ metformin , Diabex
MeSH Terms: interventions — saxagliptin

ARMS (4):
- A (Experimental): 5-mg Onglyza (saxagliptin) tablet +1000-mg Diabex extended release tablet
  Interventions: Drug: Onglyza (saxagliptin); Drug: Diabex
- B (Experimental): 5-mg saxagliptin/1000 mg metformin extended release fixed dose combination tablet
  Interventions: Drug: Onglyza (saxagliptin); Drug: 5-mg saxagliptin/1000 mg metformin
- C (Experimental): 5-mg Onglyza (saxagliptin) tablet + 500-mg Diabex extended release tablet
  Interventions: Drug: Diabex
- D (Experimental): 5-mg saxagliptin/500 mg metformin extended release fixed dose combination tablet
  Interventions: Drug: 5-mg saxagliptin/500 mg metformin

INTERVENTIONS:
Drug: Onglyza (saxagliptin) — Oral tablets, 5 mg , single dose
  Arms: A; B
Drug: Diabex — Extended release oral tablets, 1000 mg, single dose
  Arms: A
Drug: 5-mg saxagliptin/1000 mg metformin — Extended release fixed dose combination tablet, single dose
  Arms: B
Drug: Diabex — Extended release oral tablets, 500 mg, single dose
  Arms: C
Drug: 5-mg saxagliptin/500 mg metformin — Extended release fixed dose combination tablet, single dose
  Arms: D

SUMMARY:
Study in healthy subjects to measure amount of drug in blood after dosing with different saxagliptin / metformin products.

DETAILED DESCRIPTION:
Bioequivalence Study of the Fixed-dose Combination of Saxagliptin/Metformin XR Tablets Relative to Saxagliptin (Onglyza� ) Tablets and Australia-sourced Diabex XR Tablets Coadministered to Healthy Subjects in the Fed State During Steady-state Administration

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent prior to any study specific procedures
* Males or females aged 18 to 55 years (inclusive) and with a weight of at least 50 kg and a body mass index (BMI) between 18 and 35 kg/m2, inclusive
* Females must have a negative urine pregnancy test at screening and negative serum pregnancy test on admission to the unit, must not be lactating, and must be using an acceptable method of contraception for at least 1 month before dosing
* Female volunteers of childbearing potential (including perimenopausal women who have had a menstrual period within 1 year) must be using appropriate birth control (defined as a method which results in a low failure rate, ie, less than 1% per year
* Oral contraceptive and hormone replacement medications are allowed in this study if used together with a barrier contraceptive method.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate
* History or presence of gastrointestinal, hepatic, renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs (except for cholecystectomy)
* Glomerular filtration rate of less than 60 mL/min (to be estimated at screening only)
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational product (IP)
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator (eg, seasonal allergies) or history of hypersensitivity to drugs with a similar chemical structure or class to saxagliptin or metformin

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
PK Saxagliptin: Observed maximum concentration at steady state (Cmax,ss), time of maximum concentration (tmax,ss) at steady state, and area under the concentration-time curve from zero to the end of the dosing interval at steady state (AUCss) | At day 5 to day 6 at visit 2 or 3
PK : Metformin Observed maximum concentration at steady state (Cmax,ss), time of maximum concentration (tmax,ss) at steady state, and area under the concentration-time curve from zero to the end of the dosing interval at steady state (AUCss) | At day 5 to day 6 at visit 2 or 3

SECONDARY OUTCOMES:
PK : Saxagliptin 5-hydroxy Observed maximum concentration at steady state (Cmax,ss), time of maximum concentration (tmax,ss) at steady state, and area under the concentration-time curve from zero to the end of the dosing interval at steady state (AUCss) | At day 5 to day 6 at visit 2 or 3
Safety will be assessed by the incidence, severity, and relatedness of adverse events. | From day -1 visit 2 until performed follow up ( Approximately 30 days)

CONTACTS AND LOCATIONS:
Overall Officials: Miriana Kujacic, MD, Study Chair — AstraZeneca Mölndal, Sweden; Phil Leese, MD, Principal Investigator — Quintiles, Inc. Overland Park US; Peter Öhman, MD, Study Director — Astrazeneca, Wilmington, US
Locations (1):
- Research Site, Overland Park, Kansas, United States